CLINICAL TRIAL: NCT02163499
Title: Multicenter, Multi-Dose, Open-Label Maintenance of Long-Term Safety and Efficacy of Sodium Zirconium Cyclosilicate (ZS) in Hyperkalemia
Brief Title: Open-label Safety and Efficacy of Sodium Zirconium Cyclosilicate for up to 12 Months
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ZS Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ZS-005
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Results first posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-05

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia | interventions — sodium zirconium cyclosilicate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sodium Zirconium Cyclosilicate (Experimental)
  Interventions: Drug: Sodium Zirconium Cyclosilicate

INTERVENTIONS:
Drug: Sodium Zirconium Cyclosilicate — Acute Phase Dosing: Sodium Zirconium Cyclosilicate 10 g three times daily (TID) for 24 to 72 Extended Dosing: Sodium Zirconium Cyclosilicate 5 g once daily (QD). Sodium Zirconium Cyclosilicate dose increased or decreased in increments/decrements of 5 g QD up to a maximum of 15 g QD or a minimum of 5 g every other day (QOD) based on i-STAT potassium measurements up to 12 months.
  Other Names: ZS

SUMMARY:
The Open-Label Maintenance Study contains an Acute Phase, in which subjects will be dosed with ZS 10 g three times daily (tid) for 24 to 72 hours, followed by a long-term Maintenance Phase.

DETAILED DESCRIPTION:
Subjects with 2 consecutive i STAT potassium values 5.1 mmol/L will enter the Acute Phase and receive ZS 10 g tid for 24 to 72 hours, depending on potassium values. Once normokalemia (i STAT potassium between 3.5 and 5.0 mmol/L, inclusive) is restored (whether after 24, 48 or 72 hours), subjects will be enrolled in the Maintenance Phase to be dosed with ZS at a starting dose of 5 g qd. Potassium (i STAT and central laboratory) will be measured weekly throughout the first month of study and every 4 weeks thereafter through Month 12. During the Maintenance Phase, the ZS dose may be increased or decreased in increments/decrements of 5 g qd up to a maximum of 15 g qd or a minimum of 5 g every other day based on i STAT potassium measurements as outlined below:

• > 5.0 mmol/L while receiving 5 g qd or 5 g every other day or > 5.5 mmol/L while receiving 10 g qd: increase ZS dose in 5 g qd increments to a maximum dose of 15 g qd

.• Between 3.0 and 3.4 mmol/L, inclusive: decrease ZS dose in 5 g qd decrements to a minimum dose of 5 g every other day; if a subject's i STAT potassium value remains between 3.0 and 3.4 mmol/L, inclusive, on the ZS 5 g every other day dose, the subject will be withdrawn from the study and receive standard of care treatment.

There is no limit to the number of dose titrations allowed. Subjects will receive up to 12 months of treatment with open-label ZS.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent.
* Over 18 years of age.
* Two consecutive i STAT potassium values, measured 60 (+/- 15) minutes apart, both >/= 5.1 mmol/L and measured within 1 day before the first dose of ZS on Acute Phase Study Day 1.
* Ability to have repeated blood draws or effective venous catheterization.
* Women of childbearing potential must be using 2 forms of medically acceptable contraception (at least 1 barrier method) and have a negative pregnancy test at Acute Phase Study Day 1. Women who are surgically sterile or those who are postmenopausal for at least 2 years are not considered to be of childbearing potential.
* Controlled diabetic subjects.

Exclusion Criteria:

* Pseudohyperkalemia signs and symptoms, such as hemolyzed blood specimen due to excessive fist clenching to make veins prominent, difficult or traumatic venipuncture, or history of severe leukocytosis or thrombocytosis.
* Subjects treated with lactulose, rifaximin, or other non-absorbed antibiotics for hyperammonemia within 7 days prior to first dose of ZS on Acute Phase Study Day 1.
* Subjects treated with sodium polystyrene sulfonate (SPS; eg, Kayexalate®) or calcium polystyrene sulfonate (eg, Resonium®) within 3 days prior to first dose of ZS on Acute Phase Study Day 1.
* Subjects with a life expectancy of less than 12 months.
* Subjects who are severely physically or mentally incapacitated and who, in the opinion of investigator, are unable to perform the subjects' tasks associated with the protocol.
* Women who are pregnant, lactating, or planning to become pregnant.
* Subjects with diabetic ketoacidosis.
* Presence of any condition which, in the opinion of the investigator, places the subject at undue risk or potentially jeopardizes the quality of the data to be generated.
* Known hypersensitivity or previous anaphylaxis to ZS or to components thereof.
* Treatment with a drug or device within the last 30 days that has not received regulatory approval at the time of study entry.
* Subjects with cardiac arrhythmias that require immediate treatment.
* Subjects on dialysis.
* Subjects randomized into the previous ZS-002, ZS-003, ZS-004, or ZS-004E studies.
* Documented GFR <15 mL/min within 90 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 751 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Rasmussen, MD, PhD, Study Chair — ZS Pharma, Inc.
Locations (48):
- United States (34):
  - Scottsboro, Alabama
  - Tempe, Arizona
  - Tucson, Arizona
  - Chula Vista, California
  - Los Angeles, California
  - Paramount, California
  - Riverside, California
  - Sacramento, California
  - Whittier, California
  - Denver, Colorado
  - Brandon, Florida
  - DeLand, Florida
  - Hudson, Florida
  - Lauderdale Lakes, Florida
  - Miami, Florida
  - Miami Lakes, Florida
  - New Smyrna Beach, Florida
  - Tampa, Florida
  - Winter Park, Florida
  - Columbus, Georgia
  - Evergreen Park, Illinois
  - Joliet, Illinois
  - Paducah, Kentucky
  - Shreveport, Louisiana
  - Chesterfield, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Great Neck, New York
  - Providence, Rhode Island
  - Orangeburg, South Carolina
  - Sumter, South Carolina
  - Chattanooga, Tennessee
  - San Antonio, Texas
  - St. George, Utah
- Australia (5):
  - Gosford, New South Wales
  - Woolloongabba, Queensland
  - Heidelberg, Victoria
  - Melbourne, Victoria
  - Parkville, Victoria
- Germany (2):
  - Berlin
  - Stuttgart
- Amsterdam, Netherlands
- Lasi, Romania
- South Africa (4):
  - Cape Town
  - Meyerspark
  - Port Elizabeth
  - Somerset West
- Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roger SD, Lavin PT, Lerma EV, McCullough PA, Butler J, Spinowitz BS, von Haehling S, Kosiborod M, Zhao J, Fishbane S, Packham DK. Long-term safety and efficacy of sodium zirconium cyclosilicate for hyperkalaemia in patients with mild/moderate versus severe/end-stage chronic kidney disease: comparative results from an open-label, Phase 3 study. Nephrol Dial Transplant. 2021 Jan 1;36(1):137-150. doi: 10.1093/ndt/gfz285. PMID 32030422

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 56 sites in the Unites States, Australia, South Africa, Germany, the United Kingdom and the Netherlands from 23 June 2014 to 04 November 2016
Groups:
- Subject Disposition: All Screened Subjects
Period: Acute Phase: ZS 10 g TID
Arm/Group | Subject Disposition
Started | 751
Completed | 746
Not Completed | 5
Not completed — Participant's Compliance | 1
Not completed — Hypo- or Hyperkalemia | 1
Not completed — Protocol Violation | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Period: Extended Dosing Phase: ZS
Arm/Group | Subject Disposition
Started | 746
Completed | 466
Not Completed | 280
Not completed — Adverse Event | 51
Not completed — Expected Progression of CKD | 40
Not completed — Hypokalemia | 9
Not completed — Sponsor's Decision | 5
Not completed — Met ECG Withdrawal Criteria | 7
Not completed — Withdrawal by Subject | 81
Not completed — Physician Decision | 8
Not completed — Lost to Follow-up | 31
Not completed — Protocol Violation | 2
Not completed — Death | 8
Not completed — Subject Compliance | 17
Not completed — Hyperkalemia | 5
Not completed — Various reasons | 16

BASELINE CHARACTERISTICS:
Arm/Group | Acute Phase: ZS
Number analyzed (Participants) | 751
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.6 (13.03)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender Population: Acute Phase Safety Population
  Participants
    Female | 303
    Male | 448
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 25
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 89
  White | 624
  Other | 10
Use of RAAS inhibitor medication [Count of Participants; unit: Participants] — Population: Acute Phase - Safety Population
  Participants | 527
Co-morbidities at baseline [Count of Participants; unit: Participants] — Population: Acute Phase - Safety Population
  Participants
    Diabetes mellitus | 471
    Chronic kidney disease | 513
    Heart Failure | 285
Baseline eGFR [Count of Participants; unit: Participants]
  <15 | 46
  15-<30 | 243
  30-<60 | 263
  ≥60 | 190
  Missing | 9
Acute Phase baseline Serum Potassium [Count of Participants; unit: Participants] — Population: Acute Phase baseline S-K is the mean of 2 different pretreatment S-K values, recorded 60 (± 15 minutes) apart on Acute Phase Day 1.
  Participants
    <5.5 mmol/L | 287
    5.5<6.0 mmol/L | 338
    ≥6.0 mmol/L | 126

OUTCOME MEASURES:

1. Secondary Outcome: Proportion of Subjects With Mean S-K Between 3.5 and 5.5 mmol/L, Inclusive Months 3 to 12
Description: Proportion of Subjects with mean S-K between 3.5 and 5.5 mmol/L during Extended Dosing Phase - ITT Population
Time Frame: Study Days 85 to 365
Population: Extended phase ITT population
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Groups:
- Proportion: Proportion of subjects with mean S-K between 3.5 and 5.5 mmol/L, inclusive months 3 to 12
Arm/Group | Proportion
Number analyzed (Participants) | 646
Proportion of participants | 0.985 [0.972 to 0.993]

2. Secondary Outcome: Mean S-K Levels Months 3 to 12, Months 6 to 9, and Months 9 to 12.
Description: Mean S-K levels months 3 to 12(EP Days 85, 113, 141, 176, 211, 239, 267, 295, 330, 365 and EOS),months 6 to 9, and months 9 to 12.
Time Frame: Study days 85 to 365
Population: Extended phase ITT population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Mean S-K Levels Months 3 to 12,6 to 9, and 9 to 12
Number analyzed (Participants) | 734
mmol/L
  Acute Phase Baseline | 5.59 (0.425)
  Extended Dosing Days 85 to 365/End of Study: number analyzed (Participants) | 646
  Extended Dosing Days 85 to 365/End of Study | 4.66 (0.379)
  Extended Dosing Days 211 to 267: number analyzed (Participants) | 564
  Extended Dosing Days 211 to 267 | 4.68 (0.404)
  Extended Dosing Days 295 to 365: number analyzed (Participants) | 512
  Extended Dosing Days 295 to 365 | 4.62 (0.401)

3. Primary Outcome: Percent of Participants With Restoration of Normal Serum Potassium (S-K) Values (3.5 to 5.0 mmol/L, Inclusive) at the End of the Acute Phase
Description: Percentage of subjects with S-K values between 3.5 and 5.0 mmol/L, inclusive at the end of the Acute Phase - ITT Population
Time Frame: 72 Hours
Population: The Intent To Treat populations for the Acute Phase (AP-ITT) included subjects who received at least one dose of ZS with at least one S-K assessment after administration of Acute Phase ZS.
  Efficacy: Separate analyses were performed for the Acute and Extended Dosing Phases.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Percentage: Percentage of subjects with S-K values between 3.5 and 5.0 mmol/L, inclusive at the end of the Acute Phase - ITT Population
Arm/Group | Percentage
Number analyzed (Participants) | 748
Percentage of participants | 77.9 [74.8 to 80.9]

4. Primary Outcome: Percentage of Participants With Mean S-K Values ≤ 5.1 mmol/L During Extended Dosing Phase Days 85 to 365
Description: Percentage of subjects with mean S-K values ≤ 5.1 mmol/L during Extended Dosing Phase - ITT Population
Time Frame: Study Days 85 to 365
Population: The Extended Phase Intent To Treat populations (EP-ITT) included subjects who received at least one dose of ZS in the EP and have at least one S-K assessment after administration of Extended Phase ZS.
  Efficacy: Separate analyses were performed for the Acute and Extended Dosing Phases.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Percentage: Percentage of subjects with mean S-K values ≤ 5.1 mmol/L during Extended Dosing Phase - ITT Population
Arm/Group | Percentage
Number analyzed (Participants) | 646
Percentage of participants | 88.4 [85.7 to 90.8]

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | Acute Phase: ZS | Extended Dosing Phase: ZS
All-Cause Mortality (participants affected / at risk) | 0/751 | 8/746
Serious Adverse Events (participants affected / at risk) | 1/751 | 161/746
Other Adverse Events (participants affected / at risk) | 11/751 | 386/746
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Acute Phase: ZS (N=751) | Extended Dosing Phase: ZS (N=746)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 14
Cardiac failure congestive (Cardiac disorders) | 0 | 11
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Hypertension (Vascular disorders) | 0 | 4
Cellulitis (Infections and infestations) | 0 | 7
Lobar pneumonia (Infections and infestations) | 0 | 3
Acute myocardial infarction (Cardiac disorders) | 0 | 6
Fluid overload (Metabolism and nutrition disorders) | 0 | 3
Cardiac failure (Cardiac disorders) | 0 | 4
Ascites (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 3
Tropinin increased (Investigations) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Asthenia (General disorders) | 0 | 2
Ventricular tachycardia (Cardiac disorders) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 3
Osteomyelitis (Infections and infestations) | 0 | 8
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 4
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 11
Pneumonia cryptococcal (Infections and infestations) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 4
Malignant hypertension (Vascular disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Peripheral arterial occulsive disease (Vascular disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 4
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 4
Abscess limb (Infections and infestations) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Dependence on enabling machine or device (Social circumstances) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 8
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Bacteraemia (Infections and infestations) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 2
Dysarthria (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Electrocardiogram abnormal (Investigations) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hypotension (Vascular disorders) | 0 | 1
Gas gangrene (Infections and infestations) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Syncope (Nervous system disorders) | 0 | 2
Balance disorder (Nervous system disorders) | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Local swelling (General disorders) | 0 | 1
Sepsis (Infections and infestations) | 1 | 3
Appendicitis (Infections and infestations) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 3
Cardiomyopathy (Cardiac disorders) | 0 | 1
Leg amputation (Surgical and medical procedures) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 3
Multiple sclerosis (Nervous system disorders) | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Hydronephrosis (Renal and urinary disorders) | 0/746 | 1 (751)
Palpitations (Cardiac disorders) | 0 | 1
Gangrene (Infections and infestations) | 0 | 1
Necrosis (General disorders) | 0 | 1
Osteomyelitis acute (Infections and infestations) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Drug dose omission (Injury, poisoning and procedural complications) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1
Diabetic foot infection (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Heart injury (Cardiac disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pericarditis uraemic (Cardiac disorders) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Acute Phase: ZS (N=751) | Extended Dosing Phase: ZS (N=746)
Anaemia (Blood and lymphatic system disorders) | 0 | 42
Hypertension (Vascular disorders) | 1 | 78
Oedema peripheral (General disorders) | 1 | 72
Nausea (Gastrointestinal disorders) | 4 | 56
Constipation (Gastrointestinal disorders) | 2 | 46
Urinary tract infection (Infections and infestations) | 3 | 55
Upper respiratory infection (Infections and infestations) | 0 | 37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
ZS Pharma has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.